CLINICAL TRIAL: NCT03561194
Title: Omegaven Protocol:Intermediate Size Patient Population
Status: Approved for marketing | Type: Expanded Access
Sponsor: DHR Health Institute for Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 000002
Record Dates: First submitted 2018-06-04; First posted 2018-06-19 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2018-08

CONDITIONS: Parenteral Nutrition Associated Liver Disease
MeSH Terms: interventions — fish oil triglycerides

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Dietary Supplement: Omegaven — After the diagnosis of PNALD is made, patients who are followed by the Neonatal Intensive Care Unit, NICU, will contact Dr. Honrubia and Dr. Swarup. Cases may also include referrals of patients with PNALD from other healthcare facilities or self-referrals. If the patient's parents or guardians agree to participate in the study, informed consent will be obtained. The history of present illness and past medical history will be reviewed with the guardian and pertinent demographic and medical information will be recorded on data collection forms. This form will be used to record all laboratory results, nutritional history, and descriptions of any liver biopsies performed.

SUMMARY:
Children requiring prolonged courses of PN are at risk for developing PN associated liver disease. We hypothesize that although omega-6 fatty acid emulsions prevent fatty acid deficiency, they are not cleared in a manner similar to enteral chylomicrons and therefore accumulate in the liver and resulting in steatotic liver injury. We further hypothesize that a fat emulsion comprised of omega-3 fatty acids (i.e., fish oil) such as Omegaven® would be beneficial in the management of steatotic liver injury by its inhibition of de novo lipogenesis, the reduction of arachidonic acid-derived inflammatory mediators, prevention of essential fatty acid deficiency through the presence of small amounts of arachidonic acid, and improved clearance of lipids from the serum.

ELIGIBILITY:
Inclusion Criteria:

- 1. Inborn and transferred newborns born between the gestational age of 22-40 weeks who develop chronic liver failure, secondary to parenteral nutrition.

2. Patients will be PN dependent (unable to meet nutritional needs soley by enteral nutrition) and are expected to require PN for at least another 30 days 3. Patients must have diagnosis of parenteral nutrition associated liver disease (PNALD) as defined by serum direct bilirubin greater than 2mg/dL on 2 consecutive occasions 4. have had PNALD for at least four weeks prior to planned Omegaven initiation 5. Direct bilirubin > 2.0 mg/dl 6. Signed patient informed consent. 7. The patient must have utilized standard therapies to prevent the progression of his/her liver disease including surgical treatment, cyclic PN, avoiding overfeeding, reduction/removal of copper and manganese from PN, advancement of enteral feeding, and the use of ursodiol (i..e., Actigall®).

Exclusion Criteria:

- 2. Other causes of chronic liver disease (Hepatitis C, Cystic fibrosis, biliary atresia, and alpha 1 anti-trypsin deficiency,) 3. severe and/or unstable concomitant systemic disease such as complex congenital cardiac disease, renal failure, autoimmune disease, sepsis, inborn error of metabolism, genetic liver disease, 4. bleeding disorder; 5. biochemical disturbance with potential of worsening with proposed treatment, e.g. persistent hyperglycemia, hypertriglyceridemia, hypercalcemia.

6. The parent or guardian or child unwilling to provide consent or assent In rare instances, patients diagnosed with PNALD may later be found to have liver disease due to other causes in addition to the use of PN (i.e., inborn errors of metabolism, viral infections ). Such causes may not be known at the time of enrollment and will not preclude them from continuing in the study.

Ages: 22 Weeks to 40 Weeks | Sex: All
Age Groups: Child